CLINICAL TRIAL: NCT06797752
Title: Effect of the Stellate Ganglion Block on the Retinal Microcirculation: A Pilot Study
Brief Title: Effect of the Stellate Ganglion Block on the Retinal Microcirculation
Status: Recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Noah Jouett, Assistant Professor, University of Texas Southwestern Medical Center
Other Study IDs: STU-2024-1027
Record Dates: First submitted 2024-12-21; First posted 2025-01-28 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: OCTA; Severe Brain Injury; Subarachnoid Hemorrhage; Intracerebral Hemorrhage
MeSH Terms: conditions — Brain Injuries; Subarachnoid Hemorrhage; Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Intervention Group: Patients receiving the stellate ganglion block
  Interventions: Device: OCTA Scan

INTERVENTIONS:
Device: OCTA Scan — Optical Coherence Tomography Angiography before and after receiving the stellate ganglion nerve block.

SUMMARY:
Surges in the sympathetic nervous system occur at the ictus of a variety of neurological critical illnesses including intracranial hemorrhage and ischemic stroke. It is hypothesized that these exaggerated increases in sympathetic nervous activity produce maladaptations that promote secondary brain injury. One of these possible mechanisms include diffuse vasospasm that cause cerebral ischemia. Hence, methods to abrogate the sympathetic nervous system in this context are under active investigation. One possible method is the regional anesthesia technique of the stellate ganglion nerve block, which is ordinarily used for complex regional pain syndrome, but has been shown to reduce cerebral sympathetic activity and reduces vasospasm in patients with subarachnoid hemorrhage. However, its effect on the microcirculation is not clear. Hence, we propose to study patients receiving the stellate ganglion nerve block as part of their standard medical care and to image their retinal microcirculation before and after the procedure using Optical Coherence Tomography Angiography (OCTA).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Patients receiving the stellate ganglion nerve block for an approved indication, e.g. complex regional pain syndrome

Exclusion Criteria:

* Pregnancy
* Non-English speaking
* Temporary or permanent physical limitation that renders the patient unable to sit up and look inside OCTA device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving the stellate ganglion block
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-10-07 (Actual); Primary Completion 2026-10-07 (Estimated); Study Completion 2026-10-07 (Estimated)

PRIMARY OUTCOMES:
Vascular and Perfusion Density | One day
  Quantitative measure of retinal microperfusion

CONTACTS AND LOCATIONS:
Overall Officials: Noah Jouett, DO, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Pilot study

REFERENCES:
- [Background] Patton N, Aslam T, Macgillivray T, Pattie A, Deary IJ, Dhillon B. Retinal vascular image analysis as a potential screening tool for cerebrovascular disease: a rationale based on homology between cerebral and retinal microvasculatures. J Anat. 2005 Apr;206(4):319-48. doi: 10.1111/j.1469-7580.2005.00395.x. PMID 15817102